CLINICAL TRIAL: NCT04863677
Title: Effect of High-Intensity Interval Training, Moderate Continuous Training, or Guideline-Based Physical Activity on Peak Oxygen Uptake and Myocardial Fibrosis in Patients With Myocardial Infarction: Protocol for a Randomized Controlled Trial
Brief Title: The Effect of HIIT, MICT in Patients With Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Zhongshan Hospital Of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020208H(R1)
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Infarction; Cardiopulmonary Disease; Training Group, Sensitivity
Keywords: High Intensity Intermittent Training; Myocardial Infarction; Moderate Intensity Continuous Training; Cardiac Rehabilitation; Cardiopulmonary exercise testing
MeSH Terms: conditions — Myocardial Infarction; Pulmonary Heart Disease; Hypersensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Interval Training(HIIT) (Experimental): The HIIT sessions include brief, intermittent bouts of high-intensity exercise interspersed with periods of low-intensity exercise (active recovery).HIIT include 20 intervals of high-intensity (30-60s at rating of perceived exertion (RPE; Borg scale of 6-20) of 15 to 17) and low-intensity (1min at RPE <10 or totally rest). The whole exercise cycle takes around 40-50 minutes.
  Interventions: Behavioral: High Intensity Interval Training(HIIT）
- Moderate Intensity Continuous Training(MICT) (Experimental): Patients perform 40-50 minutes at a RPE of 12 to 14(a total of 4 groups, each group 5-8 min, interspersed with 2-minute rest)
  Interventions: Behavioral: Moderate Intensity Continuous Training(MICT）
- Control Group (No Intervention): No additional rehabilitation treatment or physical exercise was added in Control Group.

INTERVENTIONS:
Behavioral: High Intensity Interval Training(HIIT） — Last 12 weeks (3 sessions per week)
  Arms: High Intensity Interval Training(HIIT)
Behavioral: Moderate Intensity Continuous Training(MICT） — Moderate Intensity Continuous Training(MICT）
  Arms: Moderate Intensity Continuous Training(MICT)

SUMMARY:
This study will investigate the effect of a 12-weeks cardiac rehabilitation training (HIIT, MICT) program on VO2peak and cardiac fibrosis in patients, and evaluate the effects of HIIT on endothelial function, microvascular obstruction, body fat, inflammation, arrhythmia and psychology .

DETAILED DESCRIPTION:
Eligible and consenting patients are randomized (block randomization) in a 1:1:1 ratio. According to the number of 180 samples calculated by the sample size, the random number table containing 1-180 ( including shedding cases ) was obtained by the computer. Case number will be assigned to participants in each group according to the order of grouping, and each case number corresponded to Group1(HIIT), 2(MICT) or 3(Control) according to the random number.

The HIIT sessions include brief, intermittent bouts of high-intensity exercise interspersed with periods of low-intensity exercise (active recovery). HIIT include 20 intervals of high-intensity (30-60s at rating of perceived exertion (RPE; Borg scale of 6-20) of 15 to 17) and low-intensity (1min at RPE <10 or totally rest). The whole exercise cycle takes around 40-50 minutes (Figure 2). In MICT Group, patients perform 40-50 minutes at a RPE of 12 to 14(a total of 4 groups, each group 5-8 min, interspersed with 2-minute rest)(Figure 3). HIIT and MICT are performed only during supervised sessions with non-consecutive 3 days/week. And all patients are supervised by professional CR team. After assessing by therapists and doctors, participants also can perform three days of home-based exercises guided by wearing a sports bracelet.

The CR program includes 36 sessions supervised exercises, pharmacological counseling, patient education, catering management, smoking cessation counseling, stress management, and psychological counseling. A standard 36 sessions of CR usually lasts 12 weeks (three sessions per week).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 -75 years
2. Acute myocardial infarction (AMI) patients between 6 weeks and 3 months and had been underwent revascularization, and New York Heart Association functional classification (NYHA) Class I-III; (AMI confirmed by the World Health Organization definition (presence of symptoms of ischemia and changes in electrocardiogram) or the Third Universal Definition of Myocardial Infarction (elevation of a cardiac biomarker along with presence of either symptoms of myocardial infarction or changes in electrocardiogram))
3. Willing and able to attend the complete cardiac rehabilitation(CR)program on their own，assigned the Informed consent form.
4. Complete the cardiopulmonary exercise testing (CPET) at enrollment or has the CPET report within 1 month.

Exclusion Criteria:

1. High-intensity exercise frequently
2. Currently participating in any other clinical trials
3. Have any other diseases which limit their life to less than a year (e.g. severe valvular disease, recurrent ventricular arrhythmias, NYHA Class IV heart failure, severe aortic incompetence, severe atrial fibrillation, cancers, and end-stage renal or liver disease)
4. Dementia ; disability or sports contraindication
5. Severe acute liver failure
6. Severe acute renal failure
7. Unstable vital signs
8. Site investigators consider that the patient will be unable to complete the study and/or attend for follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
The effect of HIIT/MICT on VO2peak | 3 months
  Changes in VO2peak after 3-month cardiac rehabilitation training ( HIIT, MICT), assessed by cardiopulmonary exercise testing.
Evaluate the degree of cardiac fibrosis in 3 groups by cardiac magnetic resonance | 3 months
  The effect of HIIT/MICT on myocardial fibrosis in patients with MI, assessed by cardiac magnetic resonance.

SECONDARY OUTCOMES:
The effect of HIIT/MICT on endothelial function as assessed by the Endo-PAT2000 | 3 months
  Endothelial function will be assessed using the Endo-PAT2000 (Itamar Medical), which measures the finger pulse volume amplitude (PVA) using volume plethysmography technology to reflect peripheral blood volume changes.
The effect of HIIT/MICT on body circumference | 3 months
  The effect of HIIT/MICT on body circumference
The effect of HIIT/MICT on quality of life as assessed by SF-36 | 3 months
  The effect of HIIT/MICT on quality of life as assessed by SF-36
The effect of HIIT and MICT on depression | Baseline and 3months
  Depression is assessed by Patient Health Questionnaire - 9 (PHQ-9)
The effect of HIIT and MICT on anxiety | Baseline and 3months
  Anxiety is assessed by General anxiety disorder-7 (GAD-7)

OTHER OUTCOMES:
all-cause mortality within one year | one year
  all-cause mortality within one year
Peak oxygen uptake change | 1year, 2year and 5 year
  Changes in VO2peak after cardiac rehabilitation training ( HIIT, MICT), assessed by cardiopulmonary exercise testing.
The degree of cardiac fibrosis | 1year, 2year and 5year
  Evaluate the degree of cardiac fibrosis in 3 groups by cardiac magnetic resonance
Major adverse cardiovascular events | 1 year, 2 year and 5year
  Cardiac death, non-fatal myocardial infarction, non-fatal stroke, cardiac readmission, and revascularization
The effect of HIIT and MICT on cardiac function by MRI | Baseline and 12 weeks
  cardiac function is assessed by MRI
The effect of HIIT and MICT on other cardiopulmonary exercise testing parameters | Baseline and 12 weeks
  Other cardiopulmonary exercise testing parameters except for peak oxygen uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Qingshan Geng, Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Cardiovascular Institute, Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All data (including data dictionaries) from individuals consent to the present project, after de-identification, will be shared that include all been discussed in this article. Study protocol, statistical analysis plan, and analytic code are available for sharing. We anticipate data sharing will be ready 6 months after the publication of the primary end point of this project, and ending 36 months following article publication. Our data may be shared with investigators who provide a methodologically sound proposal with approval of an independent review committee. Proposals should be directed to gengqsh@163.net. To gain access, data requestors will need to sign a data access agreement with our institution. Data are available for 5 years at the data management center.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years

REFERENCES:
- [Derived] Shi X, Chen X, Qiu X, Luo W, Luo X, Liu H, Geng Q, Ma H, Xue L, Guo L. Effect of High-Intensity Interval Training, Moderate Continuous Training, or Guideline-Based Physical Activity on Peak Oxygen Uptake and Myocardial Fibrosis in Patients With Myocardial Infarction: Protocol for a Randomized Controlled Trial. Front Cardiovasc Med. 2022 Apr 11;9:860071. doi: 10.3389/fcvm.2022.860071. eCollection 2022. PMID 35479268